CLINICAL TRIAL: NCT00564889
Title: A Phase II Trial of Lenalidomide (Revlimid®), Cyclophosphamide and Dexamethasone in Patients With Primary Systemic Amyloidosis
Brief Title: Lenalidomide, Cyclophosphamide, and Dexamethasone in Treating Patients With Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0685; P30CA015083 (NIH); MC0685 (Other: Mayo Clinic Cancer Center); NCI-2010-01954 (Other: NCI CTRP); 06-005711 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — Cyclophosphamide; Dexamethasone; Lenalidomide

ARMS (1):
- CRD (Experimental): Lenalidomide 15mg daily (days 1-21)
  Cyclophosphamide 300 mg/m^2 (days 1, 8, 15)
  Dexamethasone 40 mg weekly
  Interventions: Drug: cyclophosphamide; Drug: dexamethasone; Drug: lenalidomide

INTERVENTIONS:
Drug: cyclophosphamide — 300 mg/m^2 days 1, 8 & 15 of a 28 day cycle taken orally with food
Drug: dexamethasone — 40 mg weekly taken orally
Drug: lenalidomide — 15 mg daily days 1-21 of a 28 day cycle taken orally with food

SUMMARY:
RATIONALE: Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop plasma cells from growing. Drugs used in chemotherapy, such as cyclophosphamide and dexamethasone, work in different ways to stop the growth of plasma cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with cyclophosphamide and dexamethasone may be an effective treatment for primary systemic amyloidosis.

PURPOSE: This phase II trial is studying how well giving lenalidomide together with cyclophosphamide and dexamethasone works in treating patients with primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the hematologic response rate in patients with primary systemic amyloidosis treated with lenalidomide, cyclophosphamide, and dexamethasone.

Secondary

* Determine the organ response rate in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the time to progression in patients treated with this regimen.
* Determine the survival of patients treated with this regimen.

OUTLINE: Patients receive oral lenalidomide on days 1-21, oral cyclophosphamide* on days 1, 8, and 15, and oral dexamethasone on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients may receive cyclophosphamide for up to 1 year. After completion of study treatment, patients are followed every 6 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histochemical diagnosis of AL amyloidosis based on detection of green birefringent material in Congo red-stained tissue specimens by polarizing microscopy
* Measurable disease, as defined by one of the following:

  * Serum monoclonal protein ≥ 1.0 g by serum electrophoresis
  * Urine monoclonal protein > 200 mg by 24-hour urine electrophoresis
  * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Symptomatic organ involvement with amyloid to justify therapy

  * May include liver involvement, cardiac involvement, renal involvement, grade 1 peripheral neuropathy, or soft tissue involvement
  * Must have more than skin purpura or carpal tunnel syndrome
* No amyloid-specific syndrome, such as carpal tunnel syndrome or skin purpura, as only evidence of disease

  - Vascular amyloid only in a bone marrow biopsy specimen or in a plasmacytoma is not indicative of systemic amyloidosis
* No clinically overt multiple myeloma (i.e., monoclonal BMPC > 30%, bone lesions, or hypercalcemia)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,000/μL
* Platelet count ≥ 75,000/μL
* Creatinine < 3.0 mg/dL
* Not pregnant
* Negative pregnancy test
* Fertile patients must use two acceptable methods of contraception for ≥ 28 days prior to, during, and for ≥ 28 days after completion of study treatment
* No nursing during and for ≥ 28 days after completion of study treatment
* No blood, semen, or sperm donation during and for ≥ 28 days after completion of study treatment
* No malignancies within the past 5 years except treated basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* No neuropathy ≥ grade 2, defined as motor neuropathy (symptomatic weakness interfering with function, but not interfering with activities of daily living [ADL]) or sensory neuropathy (sensory alteration or paresthesia [including tingling], interfering with function, but not interfering with ADL)
* No uncontrolled infection
* No syncope within the past 30 days
* No known hypersensitivity to thalidomide, including desquamating rash with thalidomide in the past
* No known seropositivity for HIV
* No active hepatitis A, B, or C
* No New York Heart Association class III or IV heart disease
* No venous thromboembolic event within the past 42 days
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation - Patients intolerant to aspirin may use low molecular weight heparin

PRIOR CONCURRENT THERAPY:

* No prior lenalidomide
* More than 2 weeks since prior and no other concurrent anticancer agents or treatments
* More than 4 weeks since prior experimental agents
* No other concurrent corticosteroids except chronic steroids (maximum dose 20 mg/day of prednisone equivalent) for disorders other than amyloidosis (e.g., adrenal insufficiency or rheumatoid arthritis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, MD, Study Chair — Mayo Clinic; Craig B. Reeder, MD, Principal Investigator — Mayo Clinic; Vivek Roy, MD, FACP, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Result] Kumar SK, Hayman SR, Buadi FK, Roy V, Lacy MQ, Gertz MA, Allred J, Laumann KM, Bergsagel LP, Dingli D, Mikhael JR, Reeder CB, Stewart AK, Zeldenrust SR, Greipp PR, Lust JA, Fonseca R, Russell SJ, Rajkumar SV, Dispenzieri A. Lenalidomide, cyclophosphamide, and dexamethasone (CRd) for light-chain amyloidosis: long-term results from a phase 2 trial. Blood. 2012 May 24;119(21):4860-7. doi: 10.1182/blood-2012-01-407791. Epub 2012 Apr 13. PMID 22504925

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-five(35) participants were recruited between December 2007 and November 2008 at Mayo Clinic.
Groups:
- Len/Cyc/Dex: Lenalidomide (Len) 15mg daily (days 1-21)
  Cyclophosphamide (Cyc) 300 mg/m^2 (days 1, 8, 15)
  Dexamethasone (Dex) 40 mg weekly
Period: Overall Study
Arm/Group | Len/Cyc/Dex
Started | 35
Completed | 6
Not Completed | 29
Not completed — Death | 7
Not completed — Adverse Event | 12
Not completed — Alternative treatment | 3
Not completed — Disease progression | 3
Not completed — Other, not specified | 4

BASELINE CHARACTERISTICS:
Groups:
- Len/Cyc/Dex: Lenalidomide (Len) 15mg daily (days 1-21); Cyclophosphamide (Cyc) 300 mg/m^2 (days 1, 8, 15); Dexamethasone (Dex) 40 mg weekly
Arm/Group | Len/Cyc/Dex
Number analyzed (Participants) | 35
Age Continuous [Median (Full Range); unit: years] | 64 [44 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 35
Received Previous Treatment [Number; unit: participants]
  Yes | 11
  No | 24
Had a Prior Stem Cell Transplant [Number; unit: participants]
  Yes | 7
  No | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Confirmed Response Defined as a Complete Response (CR), Very Good Partial Response (VGPR) or Partial Response (PR)
Description: Response that was confirmed on 2 consecutive evaluations during treatment.
  Complete Response(CR): Complete disappearance of M-protein from serum and urine on immunofixation, normalization of Free Light Chain (FLC) ratio and <5% plasma cells in bone marrow.
  Very Good Partial Response(VGPR): >=90% reduction in serum M-component; Urine M-Component <=100 mg per 24 hours.
  Partial Response(PR): >=50% reduction in serum M-component and/or Urine M-Component >=90% reduction or <200 mg per 24 hours; or >=50% decrease in difference between involved and uninvolved FLC levels.
Time Frame: Duration on study (up to 3 years)
Measure: Number; unit: participants
Arm/Group | Len/Cyc/Dex
Number analyzed (Participants) | 35
participants | 21

2. Secondary Outcome: Number of Patients With Organ Response
Description: Organ response was evaluated on the basis of improvement of one or more affected organ; only one parameter was required to satisfy the criteria. Response needed to be maintained for a minimum of 3 months to be considered valid.
  Renal response required a 50% reduction in 24-hour urine protein excretion (at least 0.5 g/d) with stable creatinine. Cardiac response required one of >= 2-mm reduction in the interventricular septal (IVS) thickness by echocardiogram, or improvement of ejection fraction by >= 20%, or improvement by 2 NYHA classes without an increase in diuretic use. Hepatic response required either >= 50% decrease in (or normalization of) an initially elevated alkaline phosphatase level or reduction in the size of the liver by at least 2 cm by radiographic determination. Gastrointestinal tract improvement was defined as normalization of a low serum carotene level, or reduction of diarrhea to < 50% of previous movements/day, or decrease in fecal fat excretion by 50%.
Time Frame: Duration of study (up to 3 years)
Measure: Number; unit: participants
Arm/Group | Len/Cyc/Dex
Number analyzed (Participants) | 35
participants | 11

3. Secondary Outcome: Number of Participants With Severe Adverse Events
Description: Severe adverse events were defined as grade 3 or higher, at least possibly related to study drugs. Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.
Time Frame: Duration of study (up to 3 years)
Measure: Number; unit: participants
Arm/Group | Len/Cyc/Dex
Number analyzed (Participants) | 35
participants | 26

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) was defined as the time from registration to hematologic progression or death of any cause. Progression free and alive patients were censored at the date of last follow-up. The median PFS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Len/Cyc/Dex
Number analyzed (Participants) | 35
months | 28.3 [12.1 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from registration to death of any cause. Surviving patients were censored at the date of last follow-up. The median OS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Len/Cyc/Dex
Number analyzed (Participants) | 35
months | 37.8 [12.3 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Groups:
- Len/Cyc/Dex: Dexamethasone (Dex) 40 mg weekly
Arm/Group | Len/Cyc/Dex
Serious Adverse Events (participants affected / at risk) | 24/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Len/Cyc/Dex (N=35)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 3 (3)
Left ventricular failure (Cardiac disorders) | 3 (4)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (2)
Intestinal necrosis (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 4 (6)
Fatigue (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 5 (6)
Urinary tract infection (Infections and infestations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 5 (5)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (3)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (4)
Confusion (Psychiatric disorders) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 3 (3)
Hemorrhage (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 6 (7)
Thrombosis (Vascular disorders) | 4 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Len/Cyc/Dex (N=35)
Hemoglobin decreased (Blood and lymphatic system disorders) | 32 (250)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 10 (17)
Hypothyroidism (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (4)
Eye disorder (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 21 (124)
Diarrhea (Gastrointestinal disorders) | 21 (90)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (2)
Enteritis (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 31 (188)
Fatigue (General disorders) | 33 (320)
Fever (General disorders) | 1 (1)
Gait abnormal (General disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 9 (11)
Sinusitis (Infections and infestations) | 3 (4)
Skin infection (Infections and infestations) | 2 (4)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 5 (5)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 15 (45)
Creatinine increased (Investigations) | 18 (156)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 29 (180)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (6)
Neutrophil count decreased (Investigations) | 21 (128)
Platelet count decreased (Investigations) | 24 (207)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (3)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (3)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (10)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 10 (56)
Memory impairment (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 9 (52)
Peripheral sensory neuropathy (Nervous system disorders) | 20 (176)
Syncope (Nervous system disorders) | 4 (6)
Anxiety (Psychiatric disorders) | 2 (3)
Depression (Psychiatric disorders) | 3 (8)
Insomnia (Psychiatric disorders) | 10 (22)
Cystitis (Renal and urinary disorders) | 6 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Rash desquamating (Skin and subcutaneous tissue disorders) | 13 (29)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes